CLINICAL TRIAL: NCT05592574
Title: Feasibility of an Il-17a Assay and Impact on Therapeutic Response in Patients With Active Axial Spondyloarthritis
Brief Title: IL17 Rate and Spondyloarthritis
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 22Rhumato02
Record Dates: First submitted 2022-10-18; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Spondylarthritis
MeSH Terms: conditions — Spondylarthritis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Spondyloarthritis without biological treatment and in failure of 2 NSAIDS
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood samples required to performe IL-17 Dosage

SUMMARY:
There are, to date, no validated biomarkers or head-to-head RCTs of biologics to guide choice of biologic agent in axSpA. While there are now two head-to-head studies of a TNF inhibitor (TNFi) vs an IL-17 inhibitor (IL-17i) in psoriatic arthritis. Recommendations refers to biological DMARDs (bDMARDs) including TNFi and IL-17i for patients with high disease activity despite the use (or intolerance/contraindication) of at least two non-steroidal anti-inflammatory drugs (NSAIDs) in axial SpA (axSpA) and in failure of a strategy including methotrexate for psoriatic arthritis. A tool to help us to decide which bDMARDs to use is necessary.

In SpA, the method of determination of IL17 seems to be questionable.

The determination of cytokines after stimulation of immune cells in patients with active SpA requiring a biological treatment could provide us with a tool to assist in the choice of therapy.

The aim of the study was to show the feasibility of cytokine assay following lymphocyte stimulation in active SpA requiring biological treatment. And secondly, to show the predictive character of this expression on the therapeutic response at three months after the implementation of a biological treatment.

ELIGIBILITY:
Inclusion criteria

* Patients with spondyloarthritis meeting the ASAS criteria
* Patients who were to benefit from the implementation of a biological treatment after failure of at least two NSAIDs.
* Patients having an active disease defined by a Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) higher than four,

Exclusion criteria

* No predominant axial manifestation,
* Having received a previous biological treatment
* Patients presenting contraindication to the implementation of these treatments.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Spondyloarthritis recruited during rheumatology consultations in rheumatology department of CHU of NICE
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2041-01-31 (Estimated); Study Completion 2041-01-31 (Estimated)

PRIMARY OUTCOMES:
to show the feasibility of cytokine assay following lymphocyte stimulation in active SpA requiring biological treatment. | 18 months
  rate of IL17

SECONDARY OUTCOMES:
predictive value of IL17 rate | 18 months
  to show the predictive character of this expression on the therapeutic response at three months after the implementation of a biological treatment. Response will be evaluated by BASDAI50

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
not schedule